CLINICAL TRIAL: NCT05280730
Title: Assessment of Neurodevelopmental Needs in Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Northwestern University (Other); University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: HM20016614
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Anonymized behavioral data and imaging data
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Boys with DMD: Boys ages 3 and above will be enrolled.
  Interventions: Other: No intervention
- Healthy boys: Healthy boys as a control group for brain imaging.

INTERVENTIONS:
Other: No intervention — There is no intervention
  Groups: Boys with DMD

SUMMARY:
Duchenne Muscular Dystrophy is a genetic disease that causes progressive muscle weakness. There is now substantial evidence that boys with this disease do not demonstrate age-related gains in their cognitive skills.

The goals of this study are (i) to use a technology-enabled neurobehavioral assessment called National Institutes of Health Toolbox Cognition Battery (NIHTB-CB) to assess brain development over time; (ii) engage with key-stakeholders to understand how neurodevelopmental problems like attention-deficit hyperactivity, autism spectrum affects individuals (and/or) families, so that we can understand meaningful effects of a potential treatment at an individual level, and (iii) to investigate using brain magnetic resonance imaging (MRI) changes in brain connectivity.

DETAILED DESCRIPTION:
Participants will be asked to do tasks such as solve puzzles, pay attention, and remember things through the NIHTB-CB administered using an IPad as well as complete questionnaires. The NIHTB-CB will be done four times (first visit, within 1 month after first visit, 12 months after first visit, and 18 months after first visit). NIHTB-CB takes about 20 to 35 minutes to complete.

Participants will also undergo brief assessment of the upper limbs; these tests will be administered by trained physical therapists and will take about 5 minutes.

Focus group: A focus group consisting of families and individuals affected by DMD will be invited to share their journey of cognitive and developmental needs. The focus group will be conducted online via the study team and is planned to last between 1 to 1.5 hours. This is optional for families.

A non-sedated brain MRI will be performed twice; scans will be separated by a one-year interval. (A child has to be age 8 or older to participate in a brain scan.) Brain imaging is optional for families.

ELIGIBILITY:
Inclusion Criteria:

* Boys with confirmed genetic mutation in the dystrophin gene
* Boys with clinical features of DMD and in whom muscle biopsy showed absence of dystrophin
* Boys with clinical features of DMD and in whom there is a family history of DMD
* Symptomatic carrier girls with DMD
* Ages 3 and above at time of study screening

Exclusion Criteria:

* Care-giver unable to give consent
* Any handicap that does not allow the ability to use an IPAD
* For MRI, braces or any metal implants.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects will be recruited nationally.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in NIHTB-CB Total Cognition Score over time | baseline and 18 months
Change in brain connectivity over time | baseline and 12 months
  Change in brain connectivity as measured by brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Mathula Thangarajh, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No